CLINICAL TRIAL: NCT06032728
Title: A Multi-site, Open, Perspective Study of Prognostic Value and Benefit From Adjuvant Targeted Therapy of Stage III Clear Cell Renal Cell Carcinoma Based on Multimodal Recurrence Scoring System
Brief Title: Multimodal Recurrence Scoring System for Stratifying Stage III Clear Cell Renal Cell Carcinoma of Receiving Adjuvant Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jun-Hang Luo, Professor, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FirstSunYatSen
Record Dates: First submitted 2023-08-30; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Renal Cell Carcinoma
Keywords: target therapy; tyrosine kinase inhibitors (TKIs)
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental): sunitinib 50 mg PO on schedule 4/2: 4 weeks on, 2 weeks off for 1 year or until disease recurrence or occurrence of a secondary malignancy, significant toxicity, or withdrawal of consent.
  Interventions: Drug: Sunitinib
- B (No Intervention): Patients with radical nephrectomy are observed without intervention

INTERVENTIONS:
Drug: Sunitinib — The investigators randomly assign multimodal recurrence scoring system defined high risk patients of stage III ccRCC into intervention group and observation group. The intervention group should receive adjuvant targeted therapy while the control group deserve observation
  Arms: A

SUMMARY:
Whether patients with stage III clear cell renal cell carcinoma (ccRCC) should receive adjuvant targeted therapy or not is still on debate. The investigators invented a multimodal recurrence scoring system that was successfully categorise patients with stage III clear cell renal cell carcinoma into high-risk and low-risk groups with Hazard Ratio (HR) of 6.21. Here the investigators randomly assign assay-defined high risk patients of locally advanced ccRCC into adjuvant targeted therapy group and observation group. Disease free survival and overall survival are the end points of observation.

ELIGIBILITY:
Inclusion Criteria:

* The informed consent has been obtained from the patient.
* With confirmed diagnosis of stage III clear cell renal cell carcinoma
* With moderate/good Eastern Cooperative Oncology Group (ECOG) health rating (PS): 0-1 score.
* The patient receive no anti-cancer treatment before primary surgery.
* The patient receive radical operation for renal cancer with negative margin.

Exclusion Criteria:

* Patients who have previously received neoadjuvant therapy
* With severe comorbidities, such as cardiovascular disease, chronic obstructive pulmonary disease, diabetes mellitus, and chronic renal dysfunction.
* With bad compliance or contraindication to enrollment.
* Pregnant woman or lactating woman.
* With contraindication to receive adjuvant targeted therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2033-10-01 (Estimated); Study Completion 2033-10-01 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | From the date of registration to up to 10 years
  Disease free survival (DFS) was defined as the time interval (in years) from the date of randomization to the first date of recurrence or occurrence of a secondary malignancy or death.

SECONDARY OUTCOMES:
Overall survival | From the date of registration to up to 10 years
  Overall survival (OS) was defined as the time from the date of randomization to the date of death due to any cause.

IPD SHARING:
Plan to Share IPD: No